CLINICAL TRIAL: NCT06080854
Title: Efficacy and Safety of AG Combined With Immunotherapy and SBRT in Patients With Potentially Resectable Pancreatic Cancer
Brief Title: AG Combined With Immunotherapy and SBRT in Patients With Potentially Resectable Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Fudan University (Other); Shanghai Changzheng Hospital (Other); The First Affiliated Hospital of Soochow University (Other); Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRAG
Record Dates: First submitted 2023-07-31; First posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-07

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — toripalimab; Gemcitabine; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Concurrent radiochemotherapy combined with immunotherapy (Experimental): Participants will receive toripalimab plus gemcitabine and nab-paclitaxel in cycles of 21 days. Non-progressors will plus concurrent radiotherapy during the 3rd cycle of chemotherapy. After 4-6 cycles treatment, Multiple disciplinary team (MDT) will evaluate whether to undergo radical surgery.
  Interventions: Drug: Toripalimab; Drug: Gemcitabine; Drug: Nab paclitaxel; Other: SBRT

INTERVENTIONS:
Drug: Toripalimab — Toripalimab 240mg administered intravenously on Days 1 of every 3 weeks
Drug: Gemcitabine — Gemcitabine 1000 mg/m^2 administered intravenously on Days 1 & 8 of every 3 weeks
Drug: Nab paclitaxel — Nab paclitaxel 125 mg/m^2 administered intravenously on Days 1 & 8 of every 3 weeks.
Other: SBRT — SBRT Radiotherapy plan: Planning gross tumor volume (PGTV) 5Gy*10 fractions, Planning target volume (PTV) 3Gy*10 fractions

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of concurrent chemoradiotherapy combined with immunotherapy in patients with potentially resectable pancreatic cancer.

DETAILED DESCRIPTION:
Due to the hidden onset and rapid progression of pancreatic cancer, most patients are already locally advanced or have distant metastasis at the time of diagnosis and lose the opportunity for surgery. Even among operable patients, about 50% will have recurrence and metastasis one year after surgery. Therefore, more and more evidence supports neoadjuvant therapy for patients with high risk factors for resectable pancreatic cancer, and conversion therapy followed by surgery for patients with borderline resectable and locally advanced pancreatic cancer. Therefore, the objective of this study is to evaluate the efficacy and safety of concurrent chemoradiotherapy combined with immunotherapy in patients with potentially resectable pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years；
2. Eastern Cooperative Oncology Group (ECOG) score of 0-1;
3. Pancreatic cancer confirmed by histology or cytology;
4. Potentially resectable pancreatic cancer documented by contrast enhanced CT (or MRI) scan;
5. Hematological indexes: Neutrophil count >= 1.5 x 10^9/L Hemoglobin >= 10g / dl Platelet count >= 100 x 10^9/L; Biochemical indicators: Total bilirubin <= 1.5 x upper limit of normal value (ULN); Aspartate aminotransferase (AST) and Alanine aminotransferase (ALT) < 1.5 x ULN; Creatinine clearance rate >= 60ml / min.
6. Participants of childbearing age need to take appropriate protective measures (contraceptive measures or other methods of birth control) before entering the group and during the test;
7. Signed informed consent;
8. Follow the protocol and follow-up procedures.

Exclusion Criteria:

1. Have received systematic anti-tumor treatment.
2. Previous history of other tumors, except for cervical cancer in situ, treated squamous cell carcinoma or bladder epithelial tumor (TA and TIS) or other malignant tumors that have received radical treatment (at least 5 years before enrollment).
3. Active bacterial or fungal infection (> = level 2 of National Cancer Institute Common Toxicity Criteria (NCI-CTC), Version 3.0).
4. Human immunodeficiency virus (HIV), hepatitis C virus (HCV), hepatitis B virus (HBV) infection, uncontrollable coronary artery disease or asthma, uncontrollable cerebrovascular disease or other diseases considered by researchers to be out of the group.
5. Autoimmune diseases or immune defects who are treated with immunosuppressive drugs.
6. Pregnant and lactating women. Pregnant women of childbearing age must be tested negative within 7 days before entering the group.
7. Drug abuse, clinical or psychological or social factors make informed consent or research implementation affected.
8. Allergic to programmed cell death protein-1 (PD-1) monoclonal antibody immunotherapy drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2025-06-06 (Estimated); Study Completion 2026-06-06 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  RECIST Version 1.1 RECIST Version 1.1 RECIST Version 1.1 RECIST Version 1.1 RECIST Version 1.1 RECIST Version 1.1
R0 resection rate | 2 years
  R0 resection rate

SECONDARY OUTCOMES:
os | 3 years
  OS is defined as the time from randomization to death due to any cause.
pfs | 3 years
  PFS is defined as the time from the first day of randomization to the date of first record of disease progression or death.
dcr | 3 years
  DCR including CR, PR, and SD
Adverse Events | 3 years
  Adverse event (AE)、Serious adverse event (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Du J, Lu C, Mao L, Zhu Y, Kong W, Shen S, Tang M, Bao S, Cheng H, Li G, Chen J, Li Q, He J, Li A, Qiu X, Gu Q, Chen D, Qi C, Song Y, Qian X, Wang L, Qiu Y, Liu B. PD-1 blockade plus chemoradiotherapy as preoperative therapy for patients with BRPC/LAPC: A biomolecular exploratory, phase II trial. Cell Rep Med. 2023 Mar 21;4(3):100972. doi: 10.1016/j.xcrm.2023.100972. Epub 2023 Mar 7. PMID 36889321